CLINICAL TRIAL: NCT01956058
Title: Recurrent Prostate Cancer After Irradiation Treated With Brachytherapy Remedial: Phase 2 Study
Brief Title: Brachytherapy for Recurrent Prostate Cancer
Acronym: CAPRICUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A01667-36
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Prostate Cancer; Brachytherapy Remedial
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- brachytherapy remedial (Experimental)
  Interventions: Radiation: brachytherapy remedial

INTERVENTIONS:
Radiation: brachytherapy remedial — brachytherapy remedial will be performed with injection of hyaluronic acid gel to interface prostate / rectum to push the rectum back and protect it from radiation.

SUMMARY:
After a curative treatment by radiotherapy for localized prostate cancer, between 20% and 50% of patients may have a biological relapse as a progressive re -rise of PSA. After prostate brachytherapy with low flow, this rate is between 2% and 6%. Depending on risk factors initially present, some patients will have a micro metastatic disease at the time of re-rise, but others will have a true local recurrence purely intra-prostate. Local recurrence after radiotherapy is associated with a high incidence of distant metastatic relapse and poor overall survival. For these reasons, the possibility of offering a local treatment for this selected population of patients can have a major therapeutic interest and allow changing a situation often considered palliative to the possibility of a second curative treatment.

Currently, there is no consensus regarding the optimal management of patients with purely local recurrence after prostate irradiation at first intention. When an external radiotherapy or brachytherapy is performed as first choice in a patient with prostate cancer, several remedial treatments have been proposed, with controversial results the decision-making for clinicians and for difficult patients. These main therapeutic options remedial (surgery, cryotherapy and brachytherapy) have the potential for complications such as rectal injury, impotence or incontinence Brachytherapy is a new salvage treatment being evaluated in the United States (Phase II study of the Radiation Therapy Oncology Group No. 0526). Several retrospective trials have shown very encouraging results in terms of acute toxicity and biochemical control in the short term. Thus, a team from Mount Sinai in New York recently published for the first time 10 years retrospective results with this approach. In their experience after treatment failures with external beam radiotherapy or brachytherapy, a dose of 122 Gy was delivered over 90% of the prostate gland. Doing this they observed biochemical control rates and survival specific of 54 % and 96 %, respectively at 10 years, with an hormone treatment associated (median 6 months) in 84 % of cases. Four patients had grade 3 toxicity or higher (11%). To reduce the rate of late toxicities the team from the University Of California San Francisco (UCSF), tested focal brachytherapy guided by functional MRI (MRI spectroscopy) to re-treat local recurrence after initial brachytherapy as monotherapy or boost. By delivering 144 Gy on recidivism objectified on MRI, the authors observed that a minimal dose of 37Gy covered 90 % of the prostate gland to treat the risk of microscopic disease. Doing this, the rate of observed toxicities and biochemical control appeared encouraging, with a median follow-up of 2 years, since no grade 3 toxicity was observed and 74% of patients achieved a PSA nadir <0.5 ng / mL without associated hormone. In case of external radiation or brachytherapy, several attempts proposed to associate an injection of hyaluronic acid gel to the prostate - rectum interface to spare healthy tissue irradiated and thus reduce the rate of radiation proctitis. The feasibility of implementing this gel has been demonstrated in patients with non- irradiated tissues. No inherent toxicity of the injection of hyaluronic acid gel has been described after prostate brachytherapy first line. The feasibility of this injection remains unproven to date on patients previously irradiated externally or by brachytherapy. We hypothesize that the risk of radiation proctitis and fistulas front prostate could be reduced using this technique in this indication.

We propose to carry out a French prospective multicenter phase II trial combining brachytherapy remedial with an injection of hyaluronic acid after surgery to reduce the risk of radiation proctitis and / or recto -urinary fistula in a patient population hyper- selected with a high probability of isolated local recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. localized prostate adenocarcinoma who presented as baseline characteristics: PSA ≤ 20ng/ml (with a rate of increase <2ng/ml/an in the 18 months preceding the biopsy diagnosis), Gleason score ≤ 7 and T1c to t2c.
2. Indication of brachytherapy remedial validated
3. Prior treatment of prostatic adenocarcinoma by radiotherapy or brachytherapy
4. Recurrence histologically proven by biopsy within ≥ 24 months after the end of the first radiotherapy or brachytherapy
5. Re-rise of PSA biochemical assays on three successive but with a PSA recurrence <10ng/ml
6. Patient over 18 years
7. WHO status 0 or 1
8. Information informed and signed by the patient or his legal representative

Exclusion Criteria:

1. Volume Prostate> 50 cm3
2. proctitis and / or radiation cystitis grade ≥ 2 at the time of inclusion
3. Initial rT3a-RT4 at the time of recurrence (clinical or MRI)
4. Gleason score ≥ 8 (if it can be established after central review) at the time of recurrence
5. lymph node and bone metastases
6. invaded the seminal vesicles (diagnosed by MRI or biopsy)
7. History of prostatectomy, TURP, or cryoablation Ablatherm ®
8. node lymphadenectomy for "restaging" before salvage treatment
9. IPSS> 12
10. Getting Started with hormone therapy since the diagnosis of recurrence
11. History of cancer within 5 years prior to entry into the trial other than basal cell skin
12. Patient already included in another clinical trial with an experimental molecule,
13. Persons deprived of liberty or under supervision (including guardianship)
14. Inability to undergo medical monitoring test for geographical, social or psychological reasons.
15. Contraindications to performing an MRI (metal prosthetic material, claustrophobia, pacemaker ...)
16. Patient anticoagulant Plavix or under
17. History of inflammatory bowel disease such as ulcerative colitis or Crohn's disease
18. History of rectal surgery

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2013-03-26 (Actual); Study Completion 2015-09-14 (Actual)

PRIMARY OUTCOMES:
Toxicity occurence | from the date of treatment up to 3 years of follow-up of the last patient treated
  The main objective of the study is to assess the occurrence of rectal and urinary toxicities grade ≥ 3 occurred within 3 years after brachytherapy remedial

SECONDARY OUTCOMES:
Investigate the observance of the injection of hyaluronic acid after surgery. | after the last treatment of the last patient in september 2015 (anticipated)
Evaluate the acute and late urinary toxicity (NCI-CTC) | for each patient from the date of the intervention up to 5 years
Assess sexual toxicities by self-administered questionnaire (IIEF 5) | for each patient every 3 months the first year following the interverntion and then evey six months up to five years
colostomy and urostomy / fistula | for each patient from the date of intervention up to the date of colostomy and / or urostomy for fistula during the follow-up period of 5 years
  The percentage of colostomy and / or urostomy for fistula and time to use a surgical procedure for patients with complications (colostomy and / or urostomy for fistula)
The time until the start of palliative hormone | for each patient from intervention date up to 5 years of follow-up
The overall survival at 5 years | for every patients from inclusion date up to five years of follow-up
Quality of life related to health EORTC QLQ C30 + EPIC survey. | for each patient every 3 months the first year following the interverntion and then evey six months up to five years
Acute and late urinary toxicity identified by self-administered questionnaire (QLQ C30 symptomatic dimensions and questionnaire scores EPIC + IPSS) | for each patient every 3 months the first year following the interverntion and then evey six months up to five years
The specific 5-year survival | from inclusion up to 5 years of follow-up for each patient
The accumulated dose delivered to the rectum after brachytherapy remedial. | after the last treatment of the last patient in september 2015 (anticipated)
survival biochemical relapse-free, according to Phoenix criteria (nadir + 2 ng/ml) | from the date of intervention up to 5 years of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre GF Leclerc, Dijon, France